CLINICAL TRIAL: NCT06513806
Title: Granisetron Versus Pethidine in Treatment of Post Spinal Shivering in Cesarean Sections
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Khaled Abdou, associated professor, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: FMASU MS84/2024
Record Dates: First submitted 2024-03-22; First posted 2024-07-22 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2024-07

CONDITIONS: Anesthesia; Adverse Effect, Spinal and Epidural
MeSH Terms: interventions — Granisetron; Meperidine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- granisetron group (Active Comparator): will receive granisetron 3 mg iv bolus
  Interventions: Drug: Granisetron 1 Mg/mL Intravenous Solution
- pethidine group (Active Comparator): will receive pethidine 25 mg iv bolus
  Interventions: Drug: Pethidin

INTERVENTIONS:
Drug: Granisetron 1 Mg/mL Intravenous Solution — will receive granisetron 3 mg iv bolus
  Arms: granisetron group
Drug: Pethidin — will receive pethidine 25 mg iv bolus
  Arms: pethidine group

SUMMARY:
Granisetron Versus Pethidine in Treatment of Post Spinal Shivering in Cesarean Sections

DETAILED DESCRIPTION:
Shivering is known to be a frequent complication, reported in 40 to 70% of patients undergoing surgery under regional anaesthesia. Shivering is a potentially serious complication, resulting in increased metabolic rate; increased oxygen consumption (up to 100-600%) along with raised carbon dioxide (CO2) production; ventilation and cardiac output; adverse postoperative outcomes.Post cesarean section spinal shivering is frequent. It causes involuntary muscular contractions and pain. Shivering, or muscular contractions, may be moderate or severe and persist for varying lengths. Anesthesia and body temperature fluctuations may produce post-spinal shivering. Properly managing post-spinal shivering improves patient outcomes and satisfaction.

Granisetron and pethidine treat post-spinal shivering. Granisetron blocks acetylcholine, a neurotransmitter that contracts muscles. Pethidine inhibits norepinephrine. Both drugs reduce post spinal shivering. However, the efficacy of granisetron and pethidine in treating post-cesarean spinal shivering has not been adequately explored.

Patients will undergo spinal anesthesia via the administration of 2.5ml of Bupivacaine 0.5% intrathecally using a 25-gauge spinal needle. The patients will be continuously monitored for any episodes of shivering, nausea, and vomiting. Vital data of the patients will also be closely monitored including oxygen saturation, pulse rate, blood pressure, respiratory rate and temperature at 10 minutes intervals throughout the operation and the stay in the recovery room. (PACU time around 30 minutes)

If shivering occurs the degree of Shivering will be classified as:

* 0: No shivering
* 1: Mild fasciculations of face or neck and ECG disturbances in the absence of voluntary activity of the arms
* 2: Visible tremor involving more than one muscle group
* 3: Gross muscular activity involving the entire body

ELIGIBILITY:
Inclusion Criteria:

* elective for caesarian section presence of post-spinal shivering, defined as involuntary muscle contractions occurring within operative and early recovery period after cesarean delivery.
* Age 18 - 45

Exclusion Criteria

* Inability to provide informed consent.
* Previous allergies or sensitivities to granisetron or pethidine.
* Current use of medications that may interact with granisetron or pethidine.
* Presence of other conditions that may contraindicate the use of granisetron or pethidine, such as known liver or kidney disease.
* Patients who are too short (<140 cm) or too tall (>190 cm)

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 330 (Actual)
Dates: Start 2024-08-01 (Actual); Primary Completion 2024-09-25 (Actual); Study Completion 2024-09-28 (Actual)

PRIMARY OUTCOMES:
treating post spinal shivering | perioperatively/periprocedurally
  If shivering occurs the degree of Shivering will be classified as:
  * 0: No shivering
  * 1: Mild fasciculations of face or neck and ECG disturbances in the absence of voluntary activity of the arms
  * 2: Visible tremor involving more than one muscle group
  * 3: Gross muscular activity involving the entire body
  assessment of tested drugs in treating post spinal shivering in patients who undergone cesarean delivery and have been treated with either granisetron or pethidine

SECONDARY OUTCOMES:
pain assessment | 12 hours postoperative
  pain scores by VAS (visual analogue scale) which is from 0-10 , 0 no Pain and 10 worst pain
nausea, vomiting | 12 hours postoperative
  incidence of postoperative complications: nausea, vomiting

CONTACTS AND LOCATIONS:
Overall Officials: Ayman M Kamaly, MD, Study Chair — Ain Shams University; David S Said, Msc, Principal Investigator — Ain Shams University
Locations (1):
- Ain Shams University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No